CLINICAL TRIAL: NCT07032493
Title: Identifying the Upper Environmental Limits of Thermal Compensation in Older Human Females Using a Rapid Humidity Ramp Protocol
Brief Title: Identifying the Limits of Survivability in Heat-exposed Older Females
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HEPRU-2025-05-A
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Heat Stress; Temperature Change, Body; Aging; Thermoregulation; Heat Exposure
Keywords: heat strain; women; heat illness; Environmental limits for compensability; heat wave; hot weather; extreme heat events
MeSH Terms: conditions — Heat Stress Disorders; Body Temperature Changes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Humidity-ramp protocol (Other): The humidity-ramp protocol will necessarily be performed first. The order of the fixed-condition exposures will be randomized.
  Interventions: Other: Humidity-Ramp Protocol
- Below-inflection fixed-condition heat exposure (5%) (Experimental): Participants will complete all exposures. The humidity-ramp protocol will necessarily be performed first. The order of the fixed-condition exposures will be randomized.
  Interventions: Other: Below-inflection fixed-condition exposure (5%)
- Control fixed-condition heat exposure (Active Comparator): Participants will complete all exposures. The humidity-ramp protocol will necessarily be performed first. The order of the fixed-condition exposures will be randomized.
  Interventions: Other: Control fixed-condition exposure
- Below-inflection fixed-condition heat exposure (10%) (Experimental): Participants will complete all exposures. The humidity-ramp protocol will necessarily be performed first. The order of the fixed-condition exposures will be randomized.
  Interventions: Other: Below-inflection fixed-condition exposure (10%)
- Above-inflection fixed-condition heat exposure (5%) (Experimental): Participants will complete all exposures. The humidity-ramp protocol will necessarily be performed first. The order of the fixed-condition exposures will be randomized.
  Interventions: Other: Above-inflection fixed-condition exposure (5%)

INTERVENTIONS:
Other: Humidity-Ramp Protocol — Participants are exposed to 42°C and 28% relative humidity for 70 minutes. Thereafter, humidity is increased 3% until an ambient humidity of 70% is achieved. The humidity at which rectal temperature inflect is subsequently determined.
  Arms: Humidity-ramp protocol
Other: Above-inflection fixed-condition exposure (5%) — After a 1 hour equilibrium at 42°C and 28% relative humidity, humidity will be increased 3% every 10 min until it is ~5% higher than the participants' rectal esophageal temperature inflection point identified in the humidity ramp protocol. These conditions will be held constant for the remainder of the 9-hour exposure period (starting from the beginning of equilibrium). Tap water will be provided at regular intervals to limit dehydration.
  Arms: Above-inflection fixed-condition heat exposure (5%)
Other: Below-inflection fixed-condition exposure (5%) — After a 1 hour equilibrium at 42°C and 28% relative humidity, humidity will be increased 3% every 10 min until it is ~5% lower than the participants' individual rectal temperature inflection point identified in the humidity ramp protocol. These conditions will be held constant for the remainder of the 9-hour exposure period (starting from the beginning of equilibrium). Tap water will be provided at regular intervals to limit dehydration.
  Arms: Below-inflection fixed-condition heat exposure (5%)
Other: Below-inflection fixed-condition exposure (10%) — After a 1 hour equilibrium at 42°C and 28% relative humidity, humidity will be increased 3% every 10 min until it is ~10% lower than the participants' individual rectal temperature inflection point identified in the humidity ramp protocol. These conditions will be held constant for the remainder of the 9-hour exposure period (starting from the beginning of equilibrium). Tap water will be provided at regular intervals to limit dehydration.
  Arms: Below-inflection fixed-condition heat exposure (10%)
Other: Control fixed-condition exposure — Participants are exposed for 9-hours to 28°C with 35% relative humidity. Participant will be allowed to drink tap water ad libitum.
  Arms: Control fixed-condition heat exposure

SUMMARY:
Climate change increases extreme heat events, elevating global heat-illness risk. Females have reduced heat loss capacity (~5%) compared to males, driven by differences in skin blood flow and sweating responses. While findings on sex-mediated mortality are mixed, some studies suggest older females (≥65 years), face higher heat-related mortality/morbidity risks, evidenced by disproportionate female deaths in the 2021 Western Heat Dome. The effects of extreme uncompensable heat on older females remain understudied.

Heat exposure initially causes net heat gain, raising core/skin temperatures and triggering heat-loss responses. Under compensable heat stress, heat loss balances gain, stabilizing core temperature. Uncompensable heat stress (exceeding maximal dissipation capacity) causes continuous core temperature rise, posing severe health risks. The specific temperature and relative humidity (RH) limits where compensability is lost are critical survival determinants, influenced by age and sex.

Ramping protocols identify these limits: participants face progressively increasing heat stress (e.g., staged humidity rises) while core temperature is monitored. Core temperature typically stabilizes initially, then exhibits an abrupt rapid increase at an inflection point, operationally defined as the limit of compensability. Despite increasing use, ramping protocol validity for accurately identifying this threshold remains unverified.

This project assesses ramping protocol validity for determining uncompensable conditions in older females and evaluates cumulative thermal and cardiovascular strain, as well as psychological and cognitive responses to both uncompensable and compensable heat. Participants will complete five trials. Trial 1 (Ramping): Rest at 42°C, 28% RH for 70min, then incremental RH increases (3% every 10min) to 70% RH. Individual core temperature (rectal) inflection points are identified from the ramping trial. Trials 2-5 (Fixed Conditions, Randomized): i) ~10% below inflection; ii) ~5% below inflection; iii) ~5% above inflection; iv) Thermo-neutral control (26°C, 45% RH). Comparing the rate of rectal temperature change and cumulative strain during prolonged fixed exposures (especially below vs. above inflection) will validate if the ramping inflection point represents the true limit of compensability for older females.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking.
* English or French speaking.
* Ability to provide informed consent.
* With or without a) chronic hypertension (elevated resting blood pressure; as defined by Heart and Stroke Canada and Hypertension Canada), b) type 2 diabetes as defined by Diabetes Canada, with at least 5 years having elapsed since time of diagnosis

Exclusion Criteria:

* Episode(s) of severe hypoglycemia (requiring the assistance of another person) within the previous year, or inability to sense hypoglycemia (hypoglycemia unawareness).
* Serious complications related to diabetes (gastroparesis, renal disease, uncontrolled hypertension, severe autonomic neuropathy).
* Uncontrolled hypertension - BP >150 mmHg systolic or >95 mmHg diastolic in a sitting position.
* Restrictions in physical activity due to disease (e.g. intermittent claudication, renal impairment, active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, severe arthritis, etc.).
* Use of or changes in medication judged by the patient or investigators to make participation in this study inadvisable.
* Cardiac abnormalities identified during screening

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Rectal temperature rate of change | End of fixed-condition heat exposure (hour 9 or termination)
  Rate of change of rectal temperature measured over the final 2-hours of heat exposure
Predicted time until 40.2°C esophageal temperature | End of fixed-condition heat exposure (hour 9 or termination)
  Estimated time for rectal temperature to reach 40.2°C, a commonly-cited criteria for severe heat-illness (e.g., heat stroke), calculated from the end-exposure rectal temperature and its rate of change (assuming this rate of change is sustained)
Core temperature (AUC) | End of fixed-condition heat exposure (hour 9 or termination)
  Area under the curve (AUC) of rectal temperature (in degree-hours) measured over the fixed-condition heat exposure

SECONDARY OUTCOMES:
Number of participants unable to finish fixed-condition heat exposure | End of fixed-condition heat exposure (hour 9 or termination)
  Number of participants who could not complete each fixed-condition heat exposure due to participant withdrawal or achieving a core temperature of 39.5°C
Mean skin temperature rate of change | End of fixed-condition heat exposure (hour 9 or termination)
  Rate of change of skin temperature measured over the final 2-hours of heat exposure
Heart rate rate of change | End of fixed-condition heat exposure (hour 9 or termination)
  Rate of change of heart rate measured over the final 2-hours of heat exposure
Heart rate (AUC) | End of fixed-condition heat exposure (hour 9 or termination)
  Area under the curve (AUC) of heart rate measured over the fixed-condition heat exposure
Thermal sensation | End of fixed-condition heat exposure (hour 9 or termination)
  Self-reported thermal sensation at the end of the fixed-condition exposures using and 8-point scale ranging from neutral (0) to extremely hot (8).
Thermal comfort | End of fixed-condition heat exposure (hour 9 or termination)
  Thermal comfort assessed via a visual analog scale ranging from extremely uncomfortable to extremely comfortable (midpoint: neutral).
Sweat rate | End of fixed-condition heat exposure (hour 9 or termination)
  Sweat rate at the end of the fixed-condition exposures (calculated via change in body weight)
Net fluid loss | End of fixed-condition heat exposure (hour 9 or termination)
  Net fluid loss estimated as the percentage change in body mass over the fixed-condition exposures.
Profiles of Mood States (POMS) | Prior to (hour 0) and at the end of fixed-condition heat exposure (hour 9 or termination)
  Potential changes in mood (7 subscales of mood: tension, anger, depression, fatigue, confusion, vigor and esteem-related affect). The POMS-40 is a validated, self-administered questionnaire that examines seven distinct aspects of mood state across two positive subscales (Esteem-Related Affect, and Vigor) and five negative subscales (Fatigue, Tension, Confusion, Anger, and Depression), which are described across 40 distinct adjectives (reference). For each individual item, participants were asked to describe "how you feel right now" by responding using a 5-point Likert scale (0 = "Not at all", 1 = "A little", 2 = "Moderately", 3 = "Quite a lot", or 4 = "Extremely"). The values of items associated with a specific subscale (e.g., Fatigue) were summed to calculate its score.
Environmental Symptoms Questionnaire (ESQ) | Prior to (hour 0) and at the end of fixed-condition heat exposure (hour 9 or termination)
  Self-reported environmental reactions and medical symptomatology associated with prolonged heat exposure. The ESQ-IV is a validated 68-item, self-administered questionnaire that has been used successfully in identifying symptomatology during exposure to a wide variety of environmental conditions, including heat exposure [24, 25]. Participants are asked to assess and described "how you have been feeling today" by responding to each item using a 6-point Likert scale (0 = "Not at all", 1 = "Slight", 2 = "Somewhat", 3 = "Moderate", 4 = "Quite a bit", or 5 = "Extreme"). Total Symptom Score was calculated from this data by taking the sum of the intensity ratings from all 68 individual items using reverse scores for the three positive items from the list ("I Felt Good", "I Felt Alert", and "I Felt Wide Awake").

OTHER OUTCOMES:
Rectal temperature inflection point | During the ramp protocol (up to 2.5 hours)
  Inflection point for rectal temperature during the humidity-ramp protocol
Heart rate inflection point | During the ramp protocol (up to 2.5 hours)
  Inflection point for heart rate during the humidity-ramp protocol

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available upon reasonable request and signed access agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available following publication of the primary study report.
Access Criteria: Reasonable request and signed access agreement